CLINICAL TRIAL: NCT03549455
Title: Augmenting Exposure Therapy With Self-Distancing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Emily Bilek, Clinical Assistant Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00141761
Record Dates: First submitted 2018-05-25; First posted 2018-06-08 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Anxiety
Keywords: anxious; anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Implosive Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exposure Therapy and Self Distancing (Experimental): All subjects will have 2 introduction sessions and then receive Exposure therapy with Self-Distancing (2 weeks) following Exposure therapy without Self-Distancing (2 weeks) followed by 2 more weeks of Exposure therapy with Self-Distancing.
  Interventions: Behavioral: Exposure Therapy and Self Distancing

INTERVENTIONS:
Behavioral: Exposure Therapy and Self Distancing — Weeks 1 and 2 will be introductory sessions (background, rationale, motivational enhancement); Weeks 3 & 4 will have Exposure therapy with Self-Distancing; Weeks 5 & 6 will have Exposure therapy only; Weeks 7 & 8 will have Exposure therapy with Self-Distancing;

SUMMARY:
Anxiety is prevalent, impairing, and costly in childhood. Evidence-based treatments for pediatric anxiety exist; however, as many as 40-60% of youth do not demonstrate optimal response. By identifying psychological factors that potentiate symptom severity and treatment response, it may be possible to strengthen these factors to treat, or even prevent the development of youth emotional disorders.

This study aims to examine whether the combination of Exposure and Self-Distancing is a feasible, acceptable, and efficient intervention for increasing perseverance in the face of exposures. This will be measured by child and parent report of treatment acceptability, examination of attendance and dropout rates, as well as participant and therapist report of participant engagement during exposures.

ELIGIBILITY:
Inclusion Criteria:

* Parent or guardian willing to give informed consent to participate
* Children who give written or oral assent
* Ages 7 and older to under 18 years old
* Has a historical anxiety diagnosis (diagnosed within the last year either within a clinical or clinical research setting) and have moderate or greater levels of current anxiety symptoms
* Current or past history of elevated symptoms of depression, obsessive-compulsive disorder and posttraumatic stress are allowable, but anxiety must be the chief complaint
* No evidence of acute risk due to suicidal intentions or behaviors in the past 6 months.

Exclusion Criteria:

* Currently receiving cognitive behavioral therapy or any other form of psychotherapy
* Have elevated symptoms of bipolar I/II disorder, schizophrenia/schizoaffective disorder, schizophreniform disorder, psychosis Not otherwise specified (NOS), mental retardation, severe behavioral concerns, or autism
* History of current substance/alcohol abuse/dependence (Past history abuse is allowable if in remission for greater than 1 year)

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2018-08-30 (Actual); Primary Completion 2020-04-09 (Actual); Study Completion 2020-04-09 (Actual)

PRIMARY OUTCOMES:
Acceptability of Self Distancing with exposure therapy | Week 8
  Treatment Acceptability Questionnaire version for the child and parent. Five Item scale (a score of 1 indicates that the care was not at all acceptable and a score of 7 would indicate a high level of acceptability). The treatment will be determined to have adequate acceptability and self-reported feasibility if parent and child report mean values greater than or equal to 5.
Feasibility of Self Distancing based on treatment completion rates | Week 8
  Total number of sessions attended. Treatment will be determined to have adequate feasibility if participants attend, on average, greater than or equal to 70% of sessions, and high feasibility if participants attend, on average greater than or equal to 80% of sessions.

SECONDARY OUTCOMES:
Treatment adherence and engagement | Weeks 3, 4, 5, 6, 7, 8
  The Treatment Engagement and Adherence Rating Scale (TEARS) will be used to assess subject completion of assigned homework, and engagement in in session practice by the child completing and therapist rating of exposure difficulty (0-10) and patient engagement (0-10).
Change in anxiety severity | Screening, Week 8
  The Screen for Childhood Anxiety-Related Emotional Disorders (SCARED) is a 41-item parent and participant-completed tool used to measure symptoms of anxiety, including the most common symptoms of panic/somatic, generalized anxiety, separation anxiety, social phobia, and school phobia. Scores range from 0-82, with higher scores indicating more severe symptoms. Both individual level changes and group mean differences will be examined.
Change in Clinical Global Impressions - Severity and improvement scale (CGI) | Screening, Weeks 1, 2, 3, 4, 5, 6, 7, 8
  This is a 2 question clinician-rated scale where the scale itself assesses overall disorder severity on a scale from 1 to 7 with 1 being "not at all" and 7 being "among the most severe cases".
Change in Clinical Global Impressions - Severity and improvement scale (CGI) | Weeks, 1, 2, 3, 4, 5, 6, 7, 8
  Only the improvement item will be completed by the parent with a score of 1 to 7 with 1 being "very much improved" and 7 being "very much worse".

CONTACTS AND LOCATIONS:
Overall Officials: Emily Bilek, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States